CLINICAL TRIAL: NCT04357002
Title: Evaluating Safety and Efficacy of Intravenous Tranexamic Acid Versus Vaginal Dinoprostone in Reducing Intraoperative Blood Loss During Abdominal Myomectomy: a Randomized Controlled Trial
Brief Title: Intravenous Tranexamic Acid Versus Vaginal Dinoprostone in Abdominal Myomectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dinoprostone tranexamic acid
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Myomectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intravenous tranexamic acid (Experimental): patients will be given a single bolus IV injection of 15 mg/kg of tranexamic acid (TXA) 20 minutes before surgical incision plus one vaginal placebo tablet 60 minutes before skin incision.
  Interventions: Drug: intravenous tranexamic acid
- vaginal dinoprostone (Active Comparator): patients will be given one vaginal dinoprostone tablet (3mg) 60 minutes before skin incision and a normal saline IV bolus 20 minutes before surgical incision
  Interventions: Drug: vaginal dinoprostone
- placebo (Placebo Comparator): patients will be given one vaginal placebo tablet 60 minutes before skin incision and a normal saline IV bolus 20 minutes before surgical incision
  Interventions: Drug: vaginal placebo

INTERVENTIONS:
Drug: intravenous tranexamic acid — patients will be given a single bolus IV injection of 15 mg/kg of tranexamic acid (TXA) 20 minutes before surgical incision plus one vaginal placebo tablet 60 minutes before skin incision.
  Arms: intravenous tranexamic acid
Drug: vaginal dinoprostone — patients will be given one vaginal dinoprostone tablet (3mg) 60 minutes before skin incision and a normal saline IV bolus 20 minutes before surgical incision
  Arms: vaginal dinoprostone
Drug: vaginal placebo — patients will be given one vaginal placebo tablet 60 minutes before skin incision and a normal saline IV bolus 20 minutes before surgical incision
  Arms: placebo

SUMMARY:
the aim of the present study is to evaluate safety and efficacy of intravenous tranexamic acid versus vaginal dinoprostone in reducing intraoperative blood loss during abdominal myomectomy

ELIGIBILITY:
Inclusion Criteria:

* symptomatic fibroids candidate for abdominal myomectomy

Exclusion Criteria:

* patients candidate for laparoscopic or hysteroscopic myomectomy or had contraindications or allergy to dinoprostone or tranexamic acid

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-04-30 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
intraoperative blood loss | one hour
  estimation of intraoperative blood loss in ml

SECONDARY OUTCOMES:
blood transfusion | 24 hours
  need for intraoperative or postoperative blood transfusion